CLINICAL TRIAL: NCT05713539
Title: Identification of the Time Taken for Skin to Return to Its Homeostatic Temperature When Exposed to Cold Conditions, and Determination of Sensitivity With Repetition
Brief Title: Determining Whether There is a Change in Time Taken to Return to Homeostatic Temperature With Repeated Exposure to a Cold Stressor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Whiteley Clinic (Other)
Responsible Party: Principal Investigator, Mark Whiteley, Consultant Venous Surgeon, The Whiteley Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TWC-MK-2022-12
Record Dates: First submitted 2023-01-25; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Needle Phobia; Needle Fear; Injection Fear
Keywords: pain; cold; skin response; injections
MeSH Terms: conditions — Iatrophobia; Pain; Common Cold

STUDY DESIGN:
Intervention Model Description: Metal placed onto skin at -2 degrees celsius for 30 seconds, and then timed on how long it takes for the skin to return to normal levels, measured using a thermal imaging camera
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cooled metal placed on skin (Experimental): Metal is placed onto the skin at a temperature of -2 degrees Celsius for 30 seconds. A thermal imaging camera will be used to identify how long it takes for the skin to return to its initial temperature.
  Interventions: Other: Metal block

INTERVENTIONS:
Other: Metal block — Small sheet of copper will be used when cooled to the designated temperature

SUMMARY:
There has been previous research suggesting cold has an effect on pain relief, however there is limited knowledge on the relationship between exposure time of a cold stressor and how long it takes to return to homeostatic temperature and normal response to cold, in addition to whether location site affects this. The skin's thermal response to a cold stimulus is not fully understood. This provides precedent for potentially using cold stressors as a way to provide pain free injections.

5 participants will be exposed to a block of copper on the skin at -2°C for 30 seconds, and a thermal camera will be used to identify the amount of time it takes for the skin to return to its homeostatic temperature. The participant will then be left for 30 seconds before the experiment is repeated to identify if there is a change in the response to cold after the first exposure.

If increased sensitivity in the response to cold occurs, the experiment will be repeated by adding an additional 30 seconds between repeats to identify the minimum time required between exposures that doesn't result in increased sensitivity. This will occur until there are two consecutive times with no increased sensitivity.

This will occur on both the forehead and on the deltoid of the arm, two areas where injections are common.

The cold stressor will be block of copper metal which will be cooled to this temperature.

DETAILED DESCRIPTION:
A thermal imaging camera is used to identify the 'normal' temperature of the skin on the forehead. A cooled block of copper is then placed onto the skin of the forehead at a temperature of -2°C for 30 seconds. A timer is then used to measure how long it takes for the skin on the forehead to return to its normal temperature. This is then repeated twice with a minute in between each measurement to identify if there is a change in the response to cold, where it takes more/less time to return to normal levels. If the time taken to return to normal changes, the participant will be given 30 minutes to rest, and then repeat the experiment with an additional minute between repeats. This will continue until there is no change in the amount of time it takes for the skin to return to normal on the forehead once exposed to the cold conditions to identify a sensitivity time due to a change in the response to cold. This will be tested on 5 patients.

This will also be tested on the outer deltoid, where injections usually occur in your arm.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed Consent
* Above 18 years old

Exclusion Criteria:

* Skin conditions or irregularities, or on medication that affects temperature regulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Measuring the time it takes to return to homeostatic temperature when exposed to cold. | 1 week
  To identify if there is sensitivity (change in response to cold) between repeats when a cold stressor when placed onto the skin which changes the amount of time it takes for the skin to return to its normal temperature

SECONDARY OUTCOMES:
To calculate the length of normal response time of skin to cold by looking at time it takes to return to homeostatic temperature in response to multiple cold exposures | 1 week
  If there is a change in response to cold, to identify how long this lasts for

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Whiteley, MS FRCS (Gen) MB BS, Principal Investigator — Executive Chairman
Locations (1):
- The Whiteley Clinic, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not planned